CLINICAL TRIAL: NCT06389032
Title: PERSEVERE in Lewy Body Dementia: A Randomized, Controlled Trial of Peer Mentor Support and Caregiver Education
Brief Title: PERSEVERE: Peer Mentor Support and Caregiver Education in Lewy Body Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jori Fleisher, Principal Investigator: Jori E Fleisher, MD MSCE, Rush University Medical Center, Department of Neurological Sciences, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21041503; 1R01AG079128-01A1 (NIH)
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Lewy Body Dementia; Parkinson Disease Dementia; Dementia With Lewy Bodies; Lewy Body Disease
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Caregiver Mentees (Experimental): Less experienced LBD family caregivers (<3 years since care recipient's cognitive impairment and/or hallucinations began) will receive PDF and website versions of the PERSEVERE modular curriculum, covering key areas of knowledge in LBD symptom and progression, caregiver strain and self-care, and links to pre-existing additional resources available on the web through various patient-facing foundations (e.g., Lewy Body Dementia Association, Parkinson's Foundation). These mentees will be matched with a trained peer mentor and will complete weekly phone or videoconference calls with each other, using the PDF and/or web-based curriculum (identical in content) as a guide for practical discussions for 12 weeks. They will complete biweekly online surveys regarding frequency, duration, and content of mentoring calls, and any falls or acute healthcare utilization of their care recipient. After the 12 weeks of mentoring, they will complete biweekly surveys for six months of follow-up.
  Interventions: Behavioral: Peer Mentor Support and Caregiver Education
- Education Group (Active Comparator): Less experienced LBD family caregivers (<3 years since care recipient's cognitive impairment and/or hallucinations began) randomized (1:1) to the education group arm will receive weekly emails from the study team delineating key topics in LBD symptom and progression, caregiver strain and self-care, and links to pre-existing additional resources available on the web through various patient-facing foundations (e.g., Lewy Body Dementia Association, Parkinson's Foundation). They will complete biweekly online surveys regarding frequency, duration, and content of mentoring calls, and any falls or acute healthcare utilization of their care recipient. After the 12 weeks of emails, they will complete biweekly surveys for six months of follow-up.
  Interventions: Behavioral: Caregiver Education
- Peer mentors (Other): Experienced LBD caregivers with >3 years' caregiving experience OR caregivers whose loved one with LBD is deceased will be recruited and trained through asynchronous and synchronous online peer mentor training to serve as mentors to less experienced LBD caregivers in the experimental arm.
  Interventions: Behavioral: Peer Mentor Support and Caregiver Education

INTERVENTIONS:
Behavioral: Peer Mentor Support and Caregiver Education — 12- week modular curriculum with handbook (PDF and Website version), additional resources and weekly phone discussions with Lewy Body Dementia (LBD) peer mentor/mentee.
  Arms: Caregiver Mentees; Peer mentors
Behavioral: Caregiver Education — 12-weeks of receiving weekly curated list of Lewy Body Dementia (LBD) educational resources based on the weekly topics via email.
  Arms: Education Group

SUMMARY:
Lewy Body Dementia (LBD) is the second most common form of degenerative dementia, affecting at least 2.4 million US adults, and the overwhelming majority of persons living with LBD (PLBD) are cared for by family caregivers. LBD caregiver strain: 1) exceeds that of non-LBD dementia caregivers; 2) worsens caregiver physical and mental health; and 3) increases the risk of PLBD hospitalization and institutionalization. LBD progression is complicated by combined motor, cognitive, and neuropsychiatric decline, and is punctuated by falls, infections, dehydration, and neuropsychiatric symptoms leading to acute healthcare utilization. Although family caregivers are uniquely positioned to identify and manage these challenges, which may avert emergency department visits and reduce morbidity, many caregivers lack the knowledge, skills, confidence, resources, and support to do so.

The study team aims to 1) quantify the impact of PERSEVERE on caregiver knowledge, attitudes, mastery, and strain; 2) identify the intervention and mentor factors determining implementation fidelity; and 3) test the effects of PERSEVERE on PLBD quality of life and healthcare utilization. This will be accomplished in an NIH Behavioral Model Stage II national, randomized, attention-controlled, 12-week trial of PERSEVERE in 502 LBD caregivers in partnership with the Lewy Body Dementia Association, Parkinson's Foundation, and LBD Caregiver Advisors. The study team will match intervention arm caregivers with a trained peer mentor who will coach them through a modular, theory-based curriculum on LBD knowledge and social support. Attention-control participants will receive weekly, curated links to educational materials. The study team will identify immediate and delayed intervention effects, including mediators of strain at 12 weeks, and caregiver strain and PLBD outcomes at nine months. Implementation fidelity and PLBD healthcare utilization will be tracked biweekly. Qualitative methods will explore the intervention- and mentor-specific factors predicting fidelity, mentee outcomes, and retention. Remote recruitment, mentoring, and community engagement strategies will maximize accessibility and inclusion of underrepresented caregiver groups. Results will illuminate the extent to which leveraging prior LBD caregivers as expert interventionists can improve current caregiver outcomes, and in turn, PLBD outcomes. These results will inform future adaptation and dissemination of this model for other conditions.

DETAILED DESCRIPTION:
Lewy body dementia (LBD) affects at least 2.4 million people in the US and is associated with cognitive, motor, and neuropsychiatric symptoms yielding higher morbidity and mortality than Alzheimer's Disease. LBD family caregiver strain: 1) exceeds that of non-LBD dementia caregivers, 2) worsens caregiver physical and mental health, and 3) independently increases the risk of hospitalization and institutionalization for persons living with LBD (PLBD). While dementia caregiver intervention research has been considerable, there has been minimal LBD caregiver research, where challenges may be greatest. PLBD have frequent emergency department (ED) visits and hospitalizations, driven by falls, infections, dehydration, and neuropsychiatric symptoms. Although family caregivers are uniquely positioned to identify and manage these challenges, which may reduce ED visits and morbidity, many caregivers lack the knowledge, skills, confidence, resources, and support to do so. NIA recognizes the gap in enhancing the knowledge and skills of dementia caregivers and the critical need to understand optimal intervention structure, content, mechanisms, and delivery methods. Without intervention, high LBD caregiver strain is associated with poorer caregiver outcomes, PLBD morbidity, and institutionalization. In non-LBD dementia and cancer, disease-specific, practical, succinct psychosocial educational interventions, and particularly those with peer mentoring-experienced caregivers coaching those earlier in the disease-have improved caregiver and patient outcomes.

The long-term goal of this work is to improve PLBD outcomes by leveraging and creating a pipeline of knowledgeable, supported family caregivers as interventionists. The overall objectives are to determine the effects of Peer Mentor Support and Caregiver Education (PERSEVERE) on LBD caregiver outcomes, define factors predicting fidelity, efficacy, and retention, and explore PLBD impact. In the PI's K23NS097615 and earlier work, the study team established the ability of a labor-intensive, interdisciplinary intervention with caregiver-focused educational materials to stabilize caregiver strain and PLBD quality of life (QoL) compared with the usual decline seen in one year. The study team then refined educational materials in a caregiver peer mentoring pilot study and documented high retention and fidelity (NIH Stage Ia).The study team has since demonstrated its ability to: 1) mitigate caregiver strain and PLBD QoL in novel interventions; 2) recruit over 200 diverse LBD caregivers in two months' time; 3) train and retain LBD caregivers as peer mentor interventionists in an NIA-funded Stage Ib study; and 4) pilot a theory-driven, peer mentor-led educational intervention yielding high retention, fidelity, satisfaction, and efficacy on key mediators of caregiver strain (knowledge, attitudes, skills, and mastery). Given prior recruitment success (achieving all of our target sample sizes in our past work), preliminary data, and longitudinal stakeholder engagement, the study team proposes an NIH Stage II (efficacy) randomized, attention-controlled trial of PERSEVERE in 502 LBD family caregivers. The study team will evaluate immediate interventional effects on mediators of caregiver strain at 12 weeks, and the delayed impact on strain, health outcomes, and PLBD six months later. The central hypothesis: Peer mentor-delivered LBD education and support will improve caregiver strain and its mediators, and PLBD health outcomes, compared with usual care. The diverse, collaborative team will use mixed methods and the RE-AIM framework to pursue the following specific aims:

Aim 1: To quantify the impact of the PERSEVERE program-an LBD-specific, peer mentor-supported educational intervention-on caregiver knowledge, attitudes, mastery, and strain.

1. Test the difference in LBD knowledge, attitudes, and mastery after 12 weeks of PERSEVERE intervention vs. attention control condition (weekly emailed resources without peer support) among LBD family caregivers.
2. Compare change in caregiver strain among active mentees vs. control caregivers at nine months.

Aim 2: To identify the intervention and peer mentor factors determining implementation fidelity.

1. Quantify the reach, adoption, implementation, and maintenance of PERSEVERE.
2. Identify matching and mentor characteristics associated with mentee outcomes and mentor retention.

Exploratory Aim 3: To test the effects of PERSEVERE on PLBD quality of life and healthcare utilization.

1. Test the difference in caregiver-reported PLBD QoL from baseline to nine months between active vs. control caregivers.
2. Quantify the difference in combined ED and hospital visits for falls, infection, dehydration, and neuropsychiatric symptoms between baseline and nine months for active and control PLBD.

ELIGIBILITY:
Inclusion Criteria:

1. Peer Mentors

   1. Participants must be 18 years of age or older.
   2. participant must be English-speaking.
   3. Participant must be US-dwelling.
   4. Participants must be either:

      1. Individuals currently cohabitating with or spending at least 10 hours weekly on caregiving for a family member diagnosed with LBD, as measured by LBCRS score ≥ 3, OR
      2. met this criterion in the past if the family member with LBD is deceased.
   5. Each participant must have access to and comfort with telephone use, including adequate hearing or appropriate assistive devices to communicate by phone.
   6. Each participant must have access to and comfort with internet use, including a working email address and adequate vision or appropriate assistive devices to be able to open and read email communications and participate in an online mentor training session.
   7. Each participant must demonstrate the capacity to consent to research participation.
   8. Each participant must not have any known terminal diagnoses or life expectancy less than 2 years, by self-report.
   9. If PLBD is alive, their cognitive or visual hallucinations have been present for 3 or more years, or between 2-3 years and caregiver actively opts for the mentor role after review of roles and responsibilities with a study team member.
2. Caregivers:

   1. Participants must be 18 years of age or older.
   2. participant must be English-speaking.
   3. Participant must be US-dwelling.
   4. Participants must be either:

      1. Individuals currently cohabitating with or spending at least 10 hours weekly on caregiving for a family member diagnosed with LBD, as measured by LBCRS score ≥ 3, OR
      2. met this criterion in the past if the family member with LBD is deceased.
   5. Caregiver must have access to and comfort with telephone use, including adequate hearing or appropriate assistive devices to communicate by phone
   6. Caregiver must have access to and comfort with internet use, including a working email address and adequate vision or appropriate assistive devices to be able to open and read email communications and participate in an online mentor training session.
   7. Caregiver must demonstrate capacity to consent to research participation.
   8. Caregiver must not have any known terminal diagnoses or life expectancy less than 2 years, by self-report
   9. PLBD cognitive symptom or visual hallucination onset within the past two years, OR symptoms for 2-3 years and after one-on-one explanation of mentor role and responsibilities with study team member, does not feel confident in ability to serve as a mentor, opts for the role of caregiver participant and being randomized to PERSEVERE or attention control.

Exclusion Criteria:

1. Peer mentors

   1. Individual is less than 18 years of age.
   2. Individual is not English-speaking.
   3. Individual is not US-dwelling.
   4. Individual who does/did not cohabitate with or spend at least 10 hours weekly on caregiving.
   5. Individual was paid for more than 50% of their caregiving responsibilities.
   6. Individual does not have access to or comfort with telephone use or lacks adequate hearing or appropriate assistive devices to communicate by phone.
   7. Individual does not have access to or comfort with internet use, including a working email address or adequate vision or appropriate assistive devices to be able to open and read email communications and participate in an online mentor training session.
   8. Individual lacks capacity to consent to research participation.
   9. PHQ-9 greater than 14, indicating severe depression.
   10. PHQ-9 question 9 (suicidal ideation) greater than 1.
   11. BGQ greater than 5, indicating complicated grief.
   12. Individual endorses a known terminal diagnosis or life expectancy less than 2 years, by self-report.
   13. PLBD cognitive symptom or visual hallucination onset less than 2 years (meeting this criterion qualifies individual as caregiver participant instead)
   14. PLBD cognitive symptom or visual hallucination onset 2-3 years ago but after one-on-one explanation of mentor role and responsibilities with study team member, does not feel confident in ability to serve as a mentor; may opt for the role of caregiver participant and being randomized to PERSEVERE or attention control.
2. Caregivers:

   1. Caregiver is less than 18 years of age.
   2. Caregiver is not English-speaking.
   3. Caregiver is not US-dwelling.
   4. Caregiver's PLBD scores 0-2 on LBCRS
   5. Caregiver does not cohabitate with or spend at least 10 hours weekly on caregiving.
   6. Caregiver is paid for more than 50% of their caregiving responsibilities.
   7. PLBD is living in a nursing facility at the time of screening.
   8. Caregiver does not have access to or comfort with telephone use, or lacks adequate hearing or appropriate assistive devices to communicate by phone.
   9. Caregiver does not have access to or comfort with internet use, including a working email address or adequate vision or appropriate assistive devices to be able to open and read email communications. and participate in an online mentor training session.
   10. PHQ-9 greater than 14, indicating severe depression.
   11. PHQ-9 question 9 (suicidal ideation) greater than 1.
   12. Caregiver lacks capacity to consent to research participation.
   13. Caregiver endorses a known terminal diagnosis or life expectancy less than 2 years, by self-report.
   14. PLBD cognitive symptoms or visual hallucinations have been present. for less than 3 years, or between 2-3 years and caregiver actively opts for the mentor role.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Caregiver Strain Index (MCSI) | Assessed at Weeks 0,12 and 38.
  An 18-item validated measurement of strain of caregiving among informal caregivers. Scores range from 0-72, with higher scores indicating higher caregiver strain.
Quality of Life in Alzheimer's Disease ( QoL-AD) | Assessed at Weeks 0, 12 and 38.
  A 13-item scale for quality of life for individuals with dementia, validated for caregiver to proxy report on person with dementia's behalf.
Dementia Attitudes Scale (DAS) | Assessed at Weeks 0,12 and 38
  A validated, 20-item scale measuring participants' attitudes toward dementia and individuals with dementia. Scores can range from 7-140, with higher scores indicating more positive attitudes
LBD Knowledge Test ( LBDK) | Assessed at Weeks 0, 12 and 38.
  A 12-item, multiple-choice test created by the study team to assess participants' level of knowledge of LBD, validated initially in a cohort of healthcare professionals (Hess SP et al, 2022). Calculated scores range from 0-100, with higher scores indicating a greater degree of knowledge of LBD and its effects.
Baseline PLBD Fall Frequency and Healthcare Utilization Questionnaire | Assessed at Week- 0 (Baseline)
  A 19-item questionnaire, developed in 2020 by PI and study team to quantify number of falls, number of healthcare utilizations, and causes of hospital encounters for a patient for whom mentees are caring. Each item scored individually, with no summary scale or total score.

SECONDARY OUTCOMES:
Fortinsky Caregiver Self-Efficacy Score | Assessed at Weeks 0, 12 and 38.
  A 9-item scale assessing two domains of caregiver self-efficacy: symptoms management self- efficacy ( items 1-5, score range 5-50) and community support services use self-efficacy (items 6-9, score range 4-40). Each item is scored using a visual analogue scale, 1-10.
Multidimensional Scale of Perceived Social Support (MSPSS) | Assessed at Weeks 0,12 and 38.
  A 12-item Likert scale scale indicating level of perceived social support by caregivers. Developed to subjectively assess the social support of an individual. Likert scale with 1 is "Very Strongly Disagree", 4 "Neutral" and 7" Very Strongly Agree"
Pearlin Mastery Scale | Assessed at Weeks 0,12 and 38
  A 7-item scale measuring the extent to which a participant sees life as being under his/her personal control vs. something that is fatalistically ruled. Score ranges from 7 to 28, with higher scores indicating greater levels of mastery

OTHER OUTCOMES:
Frequency and Duration of Mentoring Calls | Assessed at 2,4,6,8,10 and 12 weeks (Biweekly x 12 weeks)
  Online structured survey of number and duration of calls per Mentee-Mentor dyad since last survey
Study adherence of Mentors and Mentees | Assessed at Week 12 and Week 38
  Proportion of mentors and mentees dyads still in communication
Coverage of target topics; additional topics discussed | Assessed Weeks 2,4,6,8,10 and 12 weeks (Biweekly x 12 weeks)
  Online structured survey with checkboxes for topics discussed, free-text response options for additional topics.

CONTACTS AND LOCATIONS:
Overall Officials: Jori E Fleisher, MD MSCE, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No